CLINICAL TRIAL: NCT04335539
Title: A Single Arm, Open-label Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Cefiderocol in Hospitalized Paediatric Subjects 3 Months to <18 Years of Age With Suspected or Confirmed Aerobic Gram-negative Bacterial Infections
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Cefiderocol in Hospitalized Pediatric Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802R2135; 2019-002120-32 (EudraCT Number)
Expanded Access: NCT03780140 (Approved for marketing)
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Gram-negative Bacterial Infections; Bloodstream Infections (BSI); Complicated Intra-abdominal Infection (cIAI); Hospital Acquired Pneumonia (HAP); Ventilator-acquired Pneumonia; Complicated Urinary Tract Infection (cUTI); Sepsis
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Sepsis; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated | interventions — Cefiderocol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Dose Phase: Cefiderocol (Experimental): Participants will receive a single dose of cefiderocol administered intravenously (IV) on Day 1, in addition to standard of care. Participants weighing less than 34 kilograms (kg) will receive 60 milligrams (mg)/kg of cefiderocol and participants ≥34 kg will receive 2000 mg.
  Interventions: Drug: Cefiderocol; Drug: Standard of Care
- Multiple Dose Phase: Cefiderocol (Experimental): Participants will receive cefiderocol administered via IV every 8 hours on Day 1 and continuing for 5 to 14 days in addition to standard of care. Participants weighing less than 34 kg will receive 60 mg/kg of cefiderocol and participants ≥34 kg will receive 2000 mg. Dosage may be adjusted based on renal function.
  Interventions: Drug: Cefiderocol; Drug: Standard of Care

INTERVENTIONS:
Drug: Cefiderocol — Administered intravenously over 3 hours
  Other Names: S-649266; Fetroja
Drug: Standard of Care — Standard of care antibiotics will be selected by the investigator based on the suspected or confirmed pathogen(s) for the infection in accordance with local standards.

SUMMARY:
The primary objectives of this study are:

* To assess the safety and tolerability of cefiderocol after single-dose administration in hospitalized paediatric participants 3 months to < 18 years of age with suspected or confirmed aerobic Gram-negative bacterial infections
* To assess the pharmacokinetics (PK) of cefiderocol after single-dose administration of cefiderocol in hospitalized paediatric participants 3 months to < 18 years of age with suspected or confirmed aerobic Gram-negative bacterial infections
* To assess the safety and tolerability of cefiderocol after multiple-dose administration in hospitalized paediatric participants 3 months to < 12 years of age with suspected or confirmed aerobic Gram-negative bacterial infections
* To assess the PK of cefiderocol after multiple-dose administration in hospitalized paediatric participants 3 months to < 12 years of age with suspected or confirmed aerobic Gram-negative bacterial infections

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label, single- and multiple-dose study to assess the safety, tolerability, and PK of cefiderocol in hospitalized paediatric participants.

The single-dose phase will include 4 separate cohorts of participants, grouped according to age range:

* Cohort 1: 12 to < 18 years
* Cohort 2: 6 to < 12 years
* Cohort 3: 2 to < 6 years
* Cohort 4: 3 months to < 2 years Cohorts 1, 2, and 3 in the single-dose phase will be initiated in parallel. Cohort 4 will begin after safety and PK data from at least 6 participants from the single-dose Cohorts 1, 2, and 3 (with a minimum of 3 participants from Cohort 3) have been assessed.

The multiple-dose phase will include 3 cohorts according to age range (Cohorts 2, 3, and 4) and will begin after safety and PK data from 6 participants in the corresponding single-dose cohort have been assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Participant's parent(s) or legally authorized representative (LAR) provides written informed consent in accordance with regional and country-specific laws and regulations.
2. Participant provides written informed assent, when feasible (age of assent to be determined by institutional review boards/independent ethics committees [IRB's/IEC's] or be consistent with local legal requirements).
3. Hospitalized participant is 3 months to <18 years of age at the time written informed consent/assent is obtained for the single-dose phase. Hospitalized participant is 3 months to <12 years of age at the time written informed consent/assent is obtained for the multiple-dose phase. Premature babies will not be restricted, but the participant must have an adjusted or postnatal age of 3 months.
4. Participant has a suspected or confirmed infection (including but not limited to complicated urinary tract infection [cUTI], complicated intra-abdominal infection [cIAI], hospital-acquired pneumonia [HAP] /ventilator-acquired pneumonia [VAP], sepsis, or bloodstream infections [BSI]) that requires hospitalization for treatment with IV antibiotics.
5. If participant is a sexually active female of childbearing potential and has reached menarche or Tanner stage 3, participant agrees to use barrier contraception (including condom, diaphragm, or cervical cap) with spermicide or agrees to use a highly effective method of contraception (including contraceptive implant, injectable contraceptive, combination oral contraceptive, or an intrauterine [IUD] contraceptive device) from Screening up to 28 days after administration of the last dose of cefiderocol.

Exclusion Criteria:

1. Participant has a documented history of any hypersensitivity or allergic reaction to any β-lactam antibiotic (Note: for β-lactams, a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment).
2. Multiple-dose only: Participant has an infection caused only by a confirmed Gram-positive pathogen.
3. Participant has a suspected or confirmed central nervous system (CNS) infection (eg, meningitis, brain abscess, shunt infection) or osteomyelitis (which would require prolonged antibiotic therapy).
4. Participant has cystic fibrosis.
5. Single-dose phase: Participant has moderate or severe renal impairment based on estimated glomerular filtration rate (eGFR) (based on Schwartz equation if ≥ 3 months to < 1 year of age and modified Bedside Schwartz equation if ≥ 1 to < 18 years of age) of < 60 milliliter (mL) per minute (min)/1.73 ^2² at Screening.

   Multiple-dose phase: Participant has an eGFR (based on Schwartz equation if ≥ 3 months to < 1 year of age and modified Bedside Schwartz equation if ≥ 1 to < 18 years of age) of < 15 mL/min/1.73 ^2² at Screening.
6. Participant has end-stage renal disease (ESRD), is on hemodialysis (HD), or receiving continuous venovenous hemofiltration (CVVH).
7. Participant has experienced shock in the prior month or is in shock at the time of Screening.
8. Participant has severe neutropenia or is severely immunocompromised.
9. Participant has multiorgan failure.
10. Participant has a life expectancy of < 30 days due to severity of a concurrent illness.
11. Participant is a female who has a positive pregnancy test at Screening.
12. Participant is a female who is breastfeeding.
13. Participant has received any other investigational medicinal product (IMP) within 30 days.
14. Participant has any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data, including acute trauma to the pelvis or urinary tract.
15. Participant is receiving vasopressor therapy at Screening.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events in the Single Dose Phase | 28 days
Maximum Observed Plasma Concentration (Cmax) of Cefiderocol in the Single Dose Phase | Cohorts 1 and 2: Day 1 at 1, 3, 3.5, 5, and 8 hours after start of infusion. Cohorts 3 and 4: Day 1 at 3, 5, and 8 hours after the start of infusion.
Area Under the Plasma Concentration Time Curve Extrapolated From Time 0 to Infinity (AUCinf) of Cefiderocol in the Single Dose Phase | Cohorts 1 and 2: Day 1 at 1, 3, 3.5, 5, and 8 hours after start of infusion. Cohorts 3 and 4: Day 1 at 3, 5, and 8 hours after the start of infusion.
Apparent Terminal Elimination Half-life of Cefiderocol in the Single Dose Phase | Cohorts 1 and 2: Day 1 at 1, 3, 3.5, 5, and 8 hours after start of infusion. Cohorts 3 and 4: Day 1 at 3, 5, and 8 hours after the start of infusion.
Number of Participants with Adverse Events in the Multiple Dose Phase | Up to 28 days after last dose (33 to 42 days depending on treatment duration)
Maximum Observed Plasma Concentration (Cmax) of Cefiderocol in the Multiple Dose Phase | During one of the dosing intervals from the 6th to the 12th dose of cefiderocol: Cohort 2: at 1, 3, 3.5, 5, and 8 hours after start of infusion. Cohorts 3 and 4: at 3, 5, and 8 hours after start of infusion.
Area Under the Plasma Concentration Time Curve Extrapolated From Time 0 to Infinity (AUCinf) of Cefiderocol in the Multiple Dose Phase | During one of the dosing intervals from the 6th to the 12th dose of cefiderocol: Cohort 2: at 1, 3, 3.5, 5, and 8 hours after start of infusion. Cohorts 3 and 4: at 3, 5, and 8 hours after start of infusion.
Apparent Terminal Elimination Half-life of Cefiderocol in the Multiple Dose Phase | During one of the dosing intervals from the 6th to the 12th dose of cefiderocol: Cohort 2: at 1, 3, 3.5, 5, and 8 hours after start of infusion. Cohorts 3 and 4: at 3, 5, and 8 hours after start of infusion.

SECONDARY OUTCOMES:
Percentage of Participants with a Clinical Response in the Multiple Dose Phase | At 7 and 28 days after the end of treatment
Percentage of Participants with a Microbiological Response Per Pathogen in the Multiple Dose Phase | At 7 and 28 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (23):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- Estonia (2):
  - Tallinn Childrens Hospital, Tallinn
  - Tartu Ulikooli Kliinikum - Anestesioloogia ja Intensiivravi Kliinik, Tartu
- Georgia (3):
  - JSC "Medical Corporation Evex" " M. Iashvili Batumi Maternal and Child Central Hospital", Batumi
  - JSC "EVEX Medical Corporation"- M Lashvili Childrens Central Hospital, Tbilisi
  - Ltd Unimedi Kakheti Childrens New Clinic, Tbilisi
- Hungary (2):
  - Heim Pl Orszgos Gyermekgygyszati Intzet, Pilisborosjenő
  - Szegedi Tudomnyegyetem, Szegedi Tudomnyegyetem
- Latvia (2):
  - Daugavpils regional Hospital, Daugavpils
  - Bernu Kliniska Universitates Slimnica Childrens Hospital - Tornakalna, Riga
- Russia (2):
  - St. Petersburg State Pediatric Medical University, Saint Petersburg
  - Smolensk State Medical University, Smolensk
- Spain (2):
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario y Politecnico La Fe, Valencia
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Chulalongkorn University, Bangkok
  - Siriraj Hospital, Bangkok Noi
  - PHPT-Chiangrai PrachanuKroh Hospital, Chiang Mai
  - Khon Kaen University (KKU) - Faculty of Medicine-Srinagarind Hospital, Khon Kaen
- Ukraine (4):
  - Dnipropetrovsk Regional Children Clinical Hospital, Kharkiv
  - Regional Children Clinical Hospital, Kharkiv
  - National Childrens Specialized Hospital OHMATDYT of the Ministry of Health of Ukraine, Kiev
  - Higher State Educational Institute of Ukraine Ukrainian Medical Stamatological Academy, Poltava

REFERENCES:
- [Derived] Bradley JS, Orchiston E, Portsmouth S, Ariyasu M, Baba T, Katsube T, Makinde O. Pharmacokinetics, Safety and Tolerability of Single-dose or Multiple-dose Cefiderocol in Hospitalized Pediatric Patients Three Months to Less Than Eighteen Years Old With Infections Treated With Standard-of-care Antibiotics in the PEDI-CEFI Phase 2 Study. Pediatr Infect Dis J. 2025 Feb 1;44(2):136-142. doi: 10.1097/INF.0000000000004529. Epub 2024 Sep 4. PMID 39230271